CLINICAL TRIAL: NCT06786559
Title: Post Discharge Nurse-led Rehabilitation to Improve Self-care Among Stroke Patients in Bangladesh: A Pilot Randomized Controlled Trial
Brief Title: Nurse-led Rehabilitation to Improve Self-care Among Stroke Patients in Bangladesh
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hiroshima University (Other)
Responsible Party: Principal Investigator, Salma Akhter, Doctoral Researcher, Hiroshima University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 392
Record Dates: First submitted 2025-01-06; First posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Stroke; Disability Physical
Keywords: Stroke; Disability; Rehabilitation; Assistive device; Self-Care; Care Burden
MeSH Terms: conditions — Stroke; Caregiver Burden | interventions — Self-Help Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Assistive Device Intervention (Experimental): Patients and caregivers will be trained in self-care with stroke disabilities (e.g. eating, grooming, bathing, dressing, toileting), physical exercise, lifestyle modification, prevention of complications after stroke through researcher developed "Health booklet". Based on their disabilities some adjustive and exercise devices will be provided to them for improving functional independence.
  Interventions: Behavioral: Assistive Device and health Education
- Control Group (No Intervention): No "Education booklet" or adjustive device are provided to them. The patients with family caregivers in control group will receive the usual care.

INTERVENTIONS:
Behavioral: Assistive Device and health Education — After discharge they will be assessed and followed by RA nurses through home visit and tele services for 2 months. The nurses will contact the patients periodically over telephone, and follow up their regular self-care activities, adjustment to devices, exercise and adaptive behavior.
  Arms: Assistive Device Intervention

SUMMARY:
Stroke causes various levels of disability, which decreases physical function for a prolonged period. The purpose of this study is to test the feasibility and efficacy of a nurse-led rehabilitation program focused on improving the activity of daily living (ADL) among post-stroke patients in Bangladesh. A feasibility study, including descriptive and randomized controlled trial (RCT), will be conducted at the National Institute of Neuroscience & Hospital (NINS&H) in Dhaka, Bangladesh, from March 2025 to August 2025. Participants will be the post-stroke patients who got discharged from NINS&H from 5th days to 2 weeks after the onset of stroke and the family caregivers of the patients and meet the inclusion criteria. The sample size will be calculated based on G-Power analysis with a medium effect size and will be 64. The intervention will be designed to provide the 3-month nurse-led rehabilitation program regarding self-care and the use of assistive devices. Assessment for rehabilitation will be performed by the multidisciplinary team with research nurses (RA nurses), physiotherapists (PT), and occupational therapists (OT). The control group will receive the usual care. The Functional Independence Measure (FIM) measures the primary outcome as improved self-care. The secondary outcomes are self-efficacy and participation in social activities for patients and the care burden of family caregivers. We also qualitatively describe changes and improvements of cognitive, emotional, and behavioral aspects among patients and their families. The endpoints will be compared at baseline and the 3rd month. Rehabilitation with proper assistive devices may improve self-dependence, ADL, and social participation. The caregiver's burden will decrease through the implementation of self-care education and assistive devices for daily life adjustment.

DETAILED DESCRIPTION:
Stroke is considered the second most leading cause of death and disability across the globe. According to Bangladesh Sample Vital Statistics 2022, the prevalence of disability is 25.5/1000 population. Almost 70% of strokes occur in lower middle-income countries (LMICs), resulting in increased disease burden than high-income countries. Patients are often the breadwinners, and their families lose their financial footing due to treatment costs and disability, leading to economic deprivation.

Stroke rehabilitation has many barriers, including scarcity of human resources, infrastructure, finances, clinical guidelines, and national policy to support such intervention to reduce the disease burden, which is evident worldwide but much more prominent in low- and middle-income countries (LMCs). According to WHO (2019), < 10/1 million people are skilled in rehabilitation.

The purpose of this study is to test the feasibility and efficacy of nurse-assisted rehabilitation programs focused on improving the activity of daily living among post-stroke patients in Bangladesh. It can be assumed that if the nurse-assisted rehabilitation service is provided within a short time of stroke onset, the prognosis will be better, the patient will be self-dependent, the disease burden will be less, and the patient will be free of complications during post-stroke time.

A pilot randomized control trial (RCT) study will be implemented. The investigators will qualitatively and quantitatively explore the acceptance of home rehabilitation and the use of assistive devices for functional independence among post-stroke patients and their family caregivers. Investigators will also describe cognitive and emotional changes (awareness, motivation, and self-efficacy), behavior, functional changes, and social participation.

The study will be conducted at the National Institute of Neurosciences & Hospital, Dhaka, Bangladesh (NINS&H), and patients' homes. The study area is within and near the Dhaka district to reach the study participants and observe them. The study participants will be the post-stroke patients and their caregivers. The written informed consent will be taken from patients and caregivers.

The investigators will use randomized sampling techniques to select the participants. Patients who meet the inclusion criteria will be introduced by the physician at NINS&H, and research assistant (RA) nurses will contact patients and caregivers to obtain their consent. A total of 64 post-stroke patients, including 10% dropouts, will be enrolled by the researcher.

All quantitative data, including categorical data, will be described/counted/calculated with the mean with standard deviation or median and with quantile, distribution, and range. To compare feasibility and efficacy, data will be analyzed by ANOVA, ANCOVA, regression, and mixed model after checking the normality of data. Statistical significance will be set as <0.05.

The quality of the study will be assured and controlled by the Principal Investigator (PI) and other investigators. Data will be collected by the trained RA nurses.

Through participation in this study, patients and family care providers will develop comprehensive knowledge regarding stroke rehabilitation along with improved capacity of self-care activities with assistive devices. This will improve the quality of life of both stroke-affected individuals and care providers through the reduction of the caregiver's burden. The statistically significant result of this study can be disseminated to the research community of Bangladesh and to the policymakers to improve the rehabilitation facilities for long-term disabled patients with greater effort.

ELIGIBILITY:
Inclusion Criteria:

* For Patient

  1. who is 18 years old and above, both males & females,
  2. is irrespective of type of stroke and time of stroke,
  3. is within 5 days to 2 weeks of onset of the current stroke
  4. Physician advice rehabilitation, and who needs assistive devices for ADL,
  5. has family caregivers,
  6. lives in the study area, and
  7. who will provide written consent & willing to participate in the study.

For family care giver

1. Primary caregivers irrespective of sex and aged 18 years old and above, living with the patient who take care of an above patient and who meets all the inclusion criteria.
2. Who will provide written consent & willing to participate in the study

Exclusion Criteria:

* For patient

  1. Participation in other clinical trials,
  2. not having a smartphone at home, For family care giver No exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Change in the functional independence of activity of daily living | 3 months
  Functional Independence Measurement (FIM) tool will be used. This scale has 18 items from level 1-Total assistance to level 7- Complete independence. The total score is 126, the lowest score is 18. A higher score means improved functional independence level and lower score means less functional independence.

SECONDARY OUTCOMES:
Patient's Self-efficacy | 3 months
  Generalized self-efficacy scale (GSE) will be used to assess the strength of an individual's belief in oneself in difficult situations. The Scale has a total of 10 items with four-point Likert scale range from 1= not at all true to 4= Exactly true. After calculating the sum score, the total score will indicate the efficacy of participants. The lowest score is 10 & highest score is 40. Higher scores indicate higher self-efficacy.
Patient's Social participation | 3 months
  Social participation scale (short simplified) with 13 items will be used to assess the person's interaction and participation in community life as it measures the severity of social participation restrictions. The scale score ranges from 0-No restriction to 70- Extreme restriction. The higher score indicates more restriction in social participation.
Family Care burden | 3 months
  Zarit Caregiver Burden Assessment (12-items) will be used to reflect how people sometimes feel when taking care of another person. Maximum score-48, minimum score-12, higher score indicates more burden.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Laver KE, Adey-Wakeling Z, Crotty M, Lannin NA, George S, Sherrington C. Telerehabilitation services for stroke. Cochrane Database Syst Rev. 2020 Jan 31;1(1):CD010255. doi: 10.1002/14651858.CD010255.pub3. PMID 32002991
- [Background] Prvu Bettger J, Liu C, Gandhi DBC, Sylaja PN, Jayaram N, Pandian JD. Emerging Areas of Stroke Rehabilitation Research in Low- and Middle-Income Countries: A Scoping Review. Stroke. 2019 Nov;50(11):3307-3313. doi: 10.1161/STROKEAHA.119.023565. Epub 2019 Oct 17. No abstract available. PMID 31619149
- [Background] Rahman S, Sarker S, Haque AKMN, Uttsha MM, Islam MF, Deb S. AI-Driven Stroke Rehabilitation Systems and Assessment: A Systematic Review. IEEE Trans Neural Syst Rehabil Eng. 2023;31:192-207. doi: 10.1109/TNSRE.2022.3219085. Epub 2023 Jan 30. PMID 36327176
- [Background] Kim DY, Ryu B, Oh BM, Kim DY, Kim DS, Kim DY, Kim DK, Kim EJ, Lee HY, Choi H, Kim HS, Lee HH, Kim HJ, Oh HM, Seok H, Park J, Park J, Park JG, Kim JM, Lee J, Shin JH, Lee JK, Oh JS, Park KD, Kim KT, Chang MC, Chun MH, Kim MW, Kang MG, Song MK, Choi M, Ko MH, Kim NY, Paik NJ, Jung SH, Yoon SY, Lim SH, Lee SJ, Yoo SD, Lee SH, Yang SN, Park SW, Lee SY, Han SJ, Lee SJ, Bok SK, Ohn SH, Im S, Pyun SB, Hyun SE, Kim SH, Ko SH, Jee S, Kwon S, Kim TW, Chang WH, Chang WK, Yoo WK, Kim YH, Yoo YJ, Kim YW, Shin YI, Park YG, Choi YH, Kim Y; KSNR Stroke CPG Writing Group. Clinical Practice Guideline for Stroke Rehabilitation in Korea-Part 1: Rehabilitation for Motor Function (2022). Brain Neurorehabil. 2023 Jul 17;16(2):e18. doi: 10.12786/bn.2023.16.e18. eCollection 2023 Jul. PMID 37554256